CLINICAL TRIAL: NCT05476419
Title: Evaluation of Apical Gap Length and Adaptation of Custom Made Zirconia Post Using Digital Intraoral and Extraoral Scan of Conventional Silicon Impression Technique. (Randomized Controlled Clinical Trial)
Brief Title: Apical Gap Length and Adaptation of Zirconia Post Using Intraoral and Extraoral Scan of Silicon Impression Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rivan Mahmoud Gamal Mohamed El-boghdady, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Theme 3 (FPD3-3-8)RM
Record Dates: First submitted 2022-07-23; First posted 2022-07-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct intra-oral scanning technique for the post space. (Experimental): intervention will be the direct scanning of the prepared post space inside the patient mouth by using an intraoral scanner.
  Interventions: Other: Direct intra-oral scanning technique for the post space.
- In-direct scanning of the conventional post space silicone impression. (Active Comparator): The comparator will be extraoral scanning of the conventional sillicon impression of the prepared post space by using an extraoral scanner.
  Interventions: Other: Direct intra-oral scanning technique for the post space.

INTERVENTIONS:
Other: Direct intra-oral scanning technique for the post space. — scanning of prepared dental post space directly inside the patient mouth by using an intra-oral scanner

SUMMARY:
First, participants will undergo clinical and radiographic examination for taking all the needed preoperative records, then endodontically treated teeth preparation starting with removal of any carious or undermined tooth structure then ferrule preparation then followed by intra-radicular preparation and then placement of the provisional restoration. In the third visit we will take the final impression of the post space for each patient by using the intraoral scan and extraoral scan o f the conventional impression. Then assessment of the apical gap length by using digital periapical radiograph using the paralleling technique and assessment of post adaptation using replica technique followed by placement and permanent cementation of the zirconia custom made post and core restoration that showed less apical gap length and better adaptation then taking the final impression for the extracoronal restoration and finally permanent cementation of the extra coronal fixed restoration.

DETAILED DESCRIPTION:
Examination and diagnosis:Selection and examination of the patients according to inclusion and exclusion criteria. Diagnosis of the patient's chief complaint and teeth that will be involved in this study will be done.

Primary impression will be taken to produce study cast. The patients will be asked to maintain good oral hygiene measures by using tooth brush twice daily.

Taking a professional pre-operative photo.

Tooth preparation procedure:

1. Removal of any carious or undermined tooth structure then coronal preparation will be done with a ferrule of at least 1.5 to 2 mm then followed by root canal preparation to an adequate length and diameter.
2. After tooth preparation, the final impression will be taken for the post space for each participant by using the intraoral scan and extraoral scan of the conventional silicone impression.
3. Fabrication of temporary restoration using composite resin temporary material and cemented using Zinc Oxide eugenol free temporary cement.

Fabrication of restoration:

Monolithic zirconia will be used for the fabrication of post and core restoration.

Assessment of the apical gap length by using digital periapical radiograph using the paralleling technique. Assessment of post adaptation using replica technique followed by placement and permanent cementation of the zirconia custom made post and core restoration that showed less apical gap length and better adaptation. Taking the final impression for the extracoronal restoration. Finally permanent cementation of the extra coronal fixed restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-65 years with endodontically treated anterior tooth or teeth & in need of custom made post and core restoration.
2. Be physically and psychologically able to tolerate conventional restorative procedures.
3. Subject tooth free of clinical symptoms & No requirement for endodontic retreatment expressed by the presence of periapical radiolucency around an endodontically treated tooth.
4. Adequate level of oral hygiene expressed by the absence of signs of periodontal inflammation, bleeding on probing and periodontal pocket depth <4 mm.
5. Capable of signing an informed consent

Exclusion Criteria:

1. Advanced periodontitis affecting the mobility of the teeth (mobility grade II or higher)
2. Pregnant or lactating females. 3. Patients with Psychiatric problems or unrealistic expectations.

4- Patients with endodontically treated teeth which is not functioning or showing any signs or symptoms that need endodontic retreatment.

5- Occlusion problems. 6- Absence of posterior stopper.

-

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Apical gap length | through study completion, an average of 1 year".
  measuring apical gap length by the digital Periapical radiograph using the paralleling technique.

SECONDARY OUTCOMES:
Post adaptation | through study completion, an average of 1 year".
  Measuring post adaptation by using Replica technique

CONTACTS AND LOCATIONS:
Overall Officials: Rv Ma El-boghdady, Ass lecturer, Principal Investigator

IPD SHARING:
Plan to Share IPD: No